CLINICAL TRIAL: NCT01020006
Title: Phase II Study of Coagulation Factor VIIa Inhibitor PCI-27483 in Pancreatic Cancer Patients Receiving Treatment With Gemcitabine
Brief Title: Study of Safety and Tolerability of PCI-27483 in Patients With Pancreatic Cancer Patients Receiving Treatment With Gemcitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1001
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatic Cancer; Ductal Adrenocarcinoma; Exocrine Pancreatic Cancer
Keywords: PCI-27483; Factor VIIa; Gemcitabine; 4 months life expectancy; Pharmacyclics; Locally Advanced; Metastatic disease
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — PCI-27483; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine (Active Comparator): Subjects receive Gemcitabine 1000 mg/m2 weekly intravenous infusion.
  Interventions: Drug: Gemcitabine
- PCI-27483 + Gemcitabine (Experimental): Part A: Subjects received PCI-27483 0.8 mg/kg BID as initial dose and may be escalated to 1.2, and 1.5 mg/kg BID. At the same time, subjects received Gemcitabine 1000 mg/m2 weekly intravenous infusion.
  Part B: Subjects received the PCI-27483 at 1.2 mg/kg BID and Gemcitabine 1000 mg/m2 weekly intravenous infusion.
  Interventions: Drug: PCI-27483; Drug: Gemcitabine

INTERVENTIONS:
Drug: PCI-27483 — Part A: Closed to enrollment.Part B: Approximately 20 patients will be randomized to the control arm that will receive a standard regimen of gemcitabine and 20 patients will be randomized to the PCI-27483 arm and treated with both gemcitabine and PCI-27483. PCI-27483 will be administered as subcutaneous (SC) injections, nominally at a dosage of 1.2 mg/kg BID. Patients receiving PCI-27483 with a tumor response or stable disease at 12 weeks will have the option to continue PCI-27483 treatment until disease progression or the investigator considers the study treatment no longer tolerable. Treatment with gemcitabine may continue per standard of care.
  All evaluable patients will roll over into Part C at week 16 (Day 113±5). If 2 consecutive INRs at 2 hours postdose are >3.50,a reduced dosage will be calculated.
  Other Names: PCYC-1001, PCI-27483 Injection
  Arms: PCI-27483 + Gemcitabine
Drug: Gemcitabine

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of selected dose 1.2mg/kg BID dosage administered subcutaneously (SC) administered PCI-27483 to metastatic or locally advanced pancreatic cancer patients receiving concurrent therapy with intravenously administered gemcitabine for 12 weeks.

DETAILED DESCRIPTION:
This study will be conducted in three segments: Part A, Part B and Part C. Parts A and B are 12 weeks of treatment followed by 4 weeks of evaluation. In part A patients will dose-escalate up to three dose levels of PCI-27483 administered as subcutaneous (SC) injections twice-daily (BID). Part B to start once 4th patient completes 90 of 112 doses in 8 weeks. In part B patients are randomized to PCI-27483 and gemcitabine (active arm) OR gemcitabine only (control arm). PCI-27483 doses in both Part A and B will be administered in combination with a standard regimen of gemcitabine. Patients with a tumor response or stable disease at 12 weeks will have the opportunity to continue PCI-27483 treatment until disease progression or the Investigator considers the study treatment to be no longer tolerable. Treatment with gemcitabine in either the active or control arm may continue until a standard course of gemcitabine therapy has been completed. Patients will complete Part A or Part B after 16 weeks on study regardless of treatment duration. Evaluable patients will roll over into part C and be followed for 12 months from enrollment (first dose).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years old
2. Body weight ≥ 40 and ≤ 100 kg.
3. Part A: Metastatic ductal adenocarcinoma of the pancreas diagnosed ≤ 4 months prior to enrollment. (Locally advanced does not have any criteria)
4. Part B: Locally advanced ductal adenocarcinoma of the pancreas diagnosed ≤ 3 months prior to enrollment or metastatic ductal adenocarcinoma diagnosed ≤ 2 months.
5. Measurable disease by spiral CT scan (SCT) in accordance with RECIST criteria.
6. Patients after non-curative surgery are eligible if at least 4 weeks after surgery and recovered from significant surgical morbidity.
7. Estimated life expectancy of at least 4 months.
8. ECOG performance status 0 to 1.
9. Normal baseline coagulation function as defined by:

   1. PT 10-16 seconds, and
   2. aPTT 22-38 seconds.
10. Agree to not participate in contact sports or strenuous activity while taking PCI-27483.
11. Ability to understand the study, willingness to participate in the study for the study duration, and ability to provide written informed consent to participate.

Exclusion Criteria:

1. History of any clinically significant medical condition that, in the opinion of the Principal Investigator, would interfere with the study evaluation or interpretation.
2. Known history of brain metastases.
3. Any evidence of intra-cranial hemorrhage based on head CT scan within 30 days of enrollment.
4. History of disease progression while being treated with gemcitabine.
5. Radiotherapy of the primary tumor or unwillingness to defer radiotherapy of the primary tumor until > 3 months from initiation of treatment.
6. History of venous thromboembolism (eg, deep vein thrombosis, pulmonary embolism,and arterial thromboembolism) or other indications for anticoagulant treatment (eg,mechanical heart values, atrial fibrillation, etc.) within the last year. Local thrombus in the mesenteric or portal vein is acceptable.
7. Uncontrolled hypertension (systolic > 160 or diastolic > 100 mm Hg on medical treatment).
8. Continued anticoagulation therapy or anticoagulation therapy within 2 months prior to enrollment, except for perisurgical prophylaxis which must have ceased 2 weeks before enrollment.
9. Contraindication to systemic anticoagulation.
10. Continued treatment with antiplatelet drugs including aspirin, clopidogrel, etc. within the past 72 hours.
11. Known history of clinically significant or recurrent bleeding episodes, including significant bleeding after surgery, childbirth, or dental extraction.
12. Patients with documented invasion of adjacent organs by CT scan (e.g. stomach, duodenum) are not eligible
13. Patients known to have esophageal varicose are not eligible
14. Known history of a congenital coagulation factor deficiency.
15. Known acquired or hereditary platelet disorder.
16. Known history of immunodeficiency.
17. Women of child-bearing potential or sexually active men, unwilling to use adequate contraceptive protection during the course of the study.
18. Pregnant or lactating women (female patients of childbearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or if positive, pregnancy ruled out by ultrasound).
19. Laboratory Abnormalities:

    1. Serum creatinine > 2 mg/dL or creatinine clearance < 50 mL/minute (using Cockroft Gault formula)
    2. AST and ALT ≥ 4.0 x upper limit of normal (ULN).
    3. Bilirubin ≥ 3 mg/dL.
    4. Alkaline phosphatase > 5 x ULN.
    5. Albumin < 2.0g/dL.
    6. Hemoglobin < 9.0 g/dL.
    7. Platelet count < 100,000/μL.
20. Evidence of active gastrointestinal tract bleeding, including guaiac stool positivity,excluding hemorrhoidal bleeding
21. Chronic active hepatitis B or C.
22. Known HIV infection.
23. Participation in any study of an investigational device, medication, biologic, or other agent within 30 days prior to enrollment, or planned participation within the study duration.
24. Risk factors for, or use of medications known to prolong QTc interval or that may be associate with Torsades de Pointes within 7 days of treatment start (see Appendix J. Risk Factors for Drug-induced Torsades de Pointes).
25. QTc prolongation (defined as a QTc ≥ 450 msec) or other significant ECG abnormalities including 2nd degree AV block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min). If 2 screening ECGs have a QTc ≥ 450 msec, the ECGs can be submitted for a centralized, cardiologic evaluation and if determined to be < 450 msec then the patient is eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hedrick, MD, Study Director — Pharmacyclics LLC.; Laurence Elias, MD, Study Director — Pharmacyclics LLC.
Locations (17):
- United States (17):
  - TGen Clinical Reserch Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - Space Coast Medical Associates, Titusville, Florida
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Kenthucky Cancer Clinic, Hazard, Kentucky
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Beth Israel Cancer Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Summa Health System, Akron, Ohio
  - Gabrail Cancer Center Research, Canton, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - South Carolina Cancer Specialists, PA, Hilton Head, South Carolina
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - Sammons Cancer Center, Dallas, Texas
  - University of Vermont/Vermont Cancer Center, Burlington, Vermont

REFERENCES:
- See also: Related Info — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Groups:
- PCI-27483 + Gemcitabine/Part A: Part A is a nonrandomized dose escalation arm. Subjects received PCI-27483 0.8 mg/kg BID as initial dose and may be escalated to 1.2, and 1.5 mg/kg BID. At the same time, subjects received Gemcitabine 1000 mg/m2 weekly intravenous infusion on 3 out of every 4 weeks.
- PCI-27483 + Gemcitabine/Part B: Part B is a randomized arm to evaluate safety and efficacy. Subjects received PCI-27483 at 1.2 mg/kg BID and Gemcitabine 1000 mg/m2 weekly intravenous infusion.
- Gemcitabine/Part B: Subjects in this arm of Part B received Gemcitabine 1000 mg/m2 weekly intravenous infusion.
Period: Overall Study
Arm/Group | PCI-27483 + Gemcitabine/Part A | PCI-27483 + Gemcitabine/Part B | Gemcitabine/Part B
Started | 8 | 18 | 16
Completed | 0 (No subjects reached study completion as defined by protocol.) | 0 (No subjects reached study completion as defined by protocol.) | 0 (No subjects reached study completion as defined by protocol.)
Not Completed | 8 | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (PCI-27483 + Gemcitabine)/Part A | (PCI-27483 + Gemcitabine)/Part B | Gemcitabine/Part B | Total
Number analyzed (Participants) | 8 | 18 | 16 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 13 | 10 | 28
  >=65 years | 3 | 5 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 6 | 17
  Male | 4 | 11 | 10 | 25
Region of Enrollment [Number; unit: participants]
  United States | 8 | 18 | 16 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: Clinically meaningful toxicity adverse events will be defined in accordance with by CTCAE v3.0
Time Frame: First dose until 28 days after last dose of PCI-27483 or gemcitabine whichever occurs last in the assigned part (A or B).
Measure: Number; unit: participants
Arm/Group | (PCI-27483 + Gemcitabine)/Part A | (PCI-27483 + Gemcitabine)/Part B | Gemcitabine/Part B
Number analyzed (Participants) | 8 | 18 | 16
participants | 8 | 18 | 16

ADVERSE EVENTS:
Groups:
- (PCI-27483 + Gemcitabine)/Part A: Part A is a nonrandomized dose escalation arm. Subjects received PCI-27483 0.8 mg/kg BID as initial dose and may be escalated to 1.2, and 1.5 mg/kg BID. At the same time, patients received Gemcitabine 1000 mg/m2 weekly intravenous infusion on 3 out of every 4 weeks.
  All treated subjects in this group experienced at least one "treatment-emergent" adverse event.
- (PCI-27483 + Gemcitabine)/Part B: Part B is a randomized arm to evaluate safety and efficacy. Patients received PCI-27483 at 1.2 mg/kg BID and Gemcitabine 1000 mg/m2 weekly intravenous infusion.
  All treated subjects in this group experienced at least one "treatment-emergent" adverse event.
- Gemcitabine/Part B: Patients in this arm of Part B received Gemcitabine 1000 mg/m2 weekly intravenous infusion.
  All treated subjects in this group experienced at least one "treatment-emergent" adverse event.
Arm/Group | (PCI-27483 + Gemcitabine)/Part A | (PCI-27483 + Gemcitabine)/Part B | Gemcitabine/Part B
Serious Adverse Events (participants affected / at risk) | 5/8 | 12/18 | 7/16
Other Adverse Events (participants affected / at risk) | 8/8 | 18/18 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (PCI-27483 + Gemcitabine)/Part A (N=8) | (PCI-27483 + Gemcitabine)/Part B (N=18) | Gemcitabine/Part B (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (PCI-27483 + Gemcitabine)/Part A (N=8) | (PCI-27483 + Gemcitabine)/Part B (N=18) | Gemcitabine/Part B (N=16)
Anaemia (Blood and lymphatic system disorders) | 4 | 12 | 8
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 5
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 6 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 3 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 6
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5 | 5
Asthenia (General disorders) | 0 | 3 | 4
Catheter site discharge (General disorders) | 1 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 2
Early satiety (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 8 | 5
Generalised oedema (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Injection site haematoma (General disorders) | 5 | 5 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 3 | 0
Injection site reaction (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 4 | 6 | 4
Pain (General disorders) | 0 | 0 | 1
Pelvic mass (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 3
Suprapubic pain (General disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Eye infection bacterial (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine decreased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 4 | 8 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1
Platelet count increased (Investigations) | 0 | 1 | 0
Prothrombin level increased (Investigations) | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 2 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Waist circumference increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 2 | 4
White blood cell count decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 6 | 0
Drooling (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 1
Formication (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Resting tremor (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 3
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Alveolitis fibrosing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 1
Hypotension (Vascular disorders) | 1 | 0 | 2
Intra-abdominal haematoma (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No